CLINICAL TRIAL: NCT03146494
Title: The Role of Thyroid Function in the Development and Prognosis of Stanford Type A Aortic Dissection.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Beijing Anzhen Hospital
Record Dates: First submitted 2017-05-07; First posted 2017-05-10 (Actual); Last update posted 2017-05-10 (Actual); Status verified 2017-05

CONDITIONS: Stanford Type A Aortic Dissection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- STAAD
- Normal

SUMMARY:
A total of 300 consecutive cardiac patients will receive preoperative thyroid function profile evaluation, including 150 patients with Standford type A aortic dissection (STAAD) and 150 normal human.For one thing, we will compare the two groups and study the role of thyroid function in the develoment of STAAD. For another, we will collect all the perioperative data of the STAAD group and study the role of thyroid function in the prognosis of STAAD.

ELIGIBILITY:
Inclusion Criteria:

Adult patients with STAAD will underwent aortic surgery who are willing and able to give informed consent for participation in the study.

Exclusion Criteria:

The main initial exclusion criteria included clinical evidence of sepsis or cachexia or concomitant presence of any predominant severe systemic disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 300 consecutive cardiac patients will receive preoperative thyroid function profile evaluation, including 150 patients with Standford type A aortic dissection (STAAD) and 150 normal human.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2015-05-01 (Actual); Primary Completion 2017-09-01 (Estimated); Study Completion 2017-09-01 (Estimated)

PRIMARY OUTCOMES:
The Role of Thyroid Function in the Development of STAAD. | 30 days
  Patients were followed for 30-day mortality and major adverse events (MAEs) as defined by the need for rethoracotomy, occurrence of postoperative heart failure, neurologic deficit, lung failure, renal failure, or sepsis.
The Role of Thyroid Function in the Prognosis of STAAD. | 30 days
  Patients were followed for 30-day mortality and major adverse events (MAEs) as defined by the need for rethoracotomy, occurrence of postoperative heart failure, neurologic deficit, lung failure, renal failure, or sepsis.

CONTACTS AND LOCATIONS:
Locations (1):
- Wenjian Jiang, Beijing, Beijing Municipality, China